CLINICAL TRIAL: NCT05853055
Title: Disease-related Fatigue Monitoring Based on Body Signals Measured on the Skin
Acronym: Fatignals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Annaheim (Other)
Collaborators: Kliniken Valens, Klinik Gais (Unknown)
Responsible Party: Sponsor-Investigator, Simon Annaheim, Scientific Groupleader Materials-Body-Interaction Group, Empa, Swiss Federal Laboratories for Materials Science and Technology
Organization: Empa, Swiss Federal Laboratories for Materials Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5213.00284
Record Dates: First submitted 2023-03-22; First posted 2023-05-10 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Post-COVID-19 Related Fatigue
Keywords: Self-reported fatigue; Fatigue questionnaires; Continous monitoring of physiological signals; Predictive model for fatigue condition; Respiratory training
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: The study population comprises 20 patients suffering from post-COVID-19, since fatigue is a major complaint in this condition. Since abnormal breathing patterns during exertion occur mainly in post-COVID-19 patients, only these will participate in the respiratory training intervention. Half of the post-COVID-19 patients will be the control, and the other half the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-COVID-19 (respiratory training and monitoring) (Experimental): Post-COVID-19 patients allocated to this arm get an additional respiratory training added to their conventional rehabilitation program. Patients will train twice daily for the length of their rehabilitation stay. An incentive spirometer (Voldyne 5000 R, Sherwood Medical, St. Louis, USA) will be used to complete training sessions of 15 mins each.
  Interventions: Procedure: Respiratory training
- Post-COVID-19 (control and monitoring) (No Intervention): Patients receive the same therapeutical interventions as the Post-COVID19 respiratory training arm excluding respiratory training.

INTERVENTIONS:
Procedure: Respiratory training — Respiratory training will be included in the rehabilitation program of a subgroup of post-COVID-19 patients. The intervention group will train twice daily for the length of their rehabilitation stay using an incentive spirometer (Voldyne 5000 R, Sherwood Medical, St. Louis, USA). Subjects will be instructed to first completely exhale slowly. Then inspire slowly up to 70% of their vital capacity, producing a constant flow controlled via feedback from the device. This procedure will be repeated every 30 s (paced by a metronome) for 15 min. The training will be conducted twice a day, resulting in a total of 60 inspirations per day.
  Arms: Post-COVID-19 (respiratory training and monitoring)

SUMMARY:
This study investigates the use of physiological parameters as predictors of disease-related fatigue. For that purpose, wearable devices are used to monitor post-COVID-19 patients during their stay in a rehabilitation clinic. Besides, the effectiveness of respiratory training in reducing breathlessness and improving exercise breathing patterns in patients suffering from post-COVID-19 will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* suffering from post-COVID-19 fatigue (i.e., score equal or higher than 5 on the single-item fatigue [SIF] or the Fatigue Severity Scale [FSS])
* admitted to Gais rehabilitation clinic
* able to use a mobile phone
* able to wear and handle the monitoring devices

Exclusion Criteria:

* Patients suffering from a relevant comorbidity (i.e., comorbidity resulting in significant distortion of physiological signals [e.g., moderate to severe chronic obstructive pulmonary disease or persistent atrial fibrillation])
* pregnancy
* unable to use, wear or handle the monitoring systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Quantification of fatigue based on self-reported fatigue by means of single item fatigue questionnaire | baseline
  The single item fatigue (SIF) questionnaire is a multidimensional questionnaire developed for use in daily clinical practice. It has 5-items covering global fatigue, cognitive fatigue, emotional fatigue, physical fatigue, fatigue relief by sleep), each consisting of an 11-point likert scale (0 [no fatigue] to 10 [severe fatigue]), . Perceived fatigue was asked for the past 24 hours.
Quantification of fatigue based on self-reported fatigue by means of single item fatigue questionnaire | after 12 weeks of rehabilitation
  The single item fatigue (SIF) questionnaire is a multidimensional questionnaire developed for use in daily clinical practice. It has 5-items covering global fatigue, cognitive fatigue, emotional fatigue, physical fatigue, fatigue relief by sleep), each consisting of an 11-point likert scale (0 [no fatigue] to 10 [severe fatigue]), . Perceived fatigue was asked for the past 24 hours.
Heart rate | baseline
  Heart rate (in beats per minute) will be obtained from ECG signals monitored continuously by the eqO2+ LifeMonitor (Equivital Inc, New York, USA)
Heart rate | after 12 weeks of rehabilitation
  Heart rate (in beats per minute) will be obtained from ECG signals monitored continuously by the eqO2+ LifeMonitor (Equivital Inc, New York, USA)
Heart rate variability | baseline
  Heart rate variability (in milliseconds) will be obtained from ECG signals monitored continuously by the eqO2+ LifeMonitor (Equivital Inc, New York, USA)
Heart rate variability | after 12 weeks of rehabilitation
  Heart rate variability (in milliseconds) will be obtained from ECG signals monitored continuously by the eqO2+ LifeMonitor (Equivital Inc, New York, USA)
Breathing rate | baseline
  Breathing rate (in breaths per minute) will be obtained from breathing waveform signals monitored continuously by the eqO2+ LifeMonitor (Equivital Inc, New York, USA)
Breathing rate | after 12 weeks of rehabilitation
  Breathing rate (in breaths per minute) will be obtained from breathing waveform signals monitored continuously by the eqO2+ LifeMonitor (Equivital Inc, New York, USA)
Physical activity intensity | baseline
  The mean amplitude observed for the resultant acceleration (based on 3D acceleration measurements in g) is considered to be representative for the physical activity intensity. It will be obtained from acceleration measurements monitored continuously by the eqO2+ LifeMonitor (Equivital Inc, New York, USA)
Physical activity intensity | after 12 weeks of rehabilitation
  The mean amplitude observed for the resultant acceleration (based on 3D acceleration measurements in g) is considered to be representative for the physical activity intensity. It will be obtained from acceleration measurements monitored continuously by the eqO2+ LifeMonitor (Equivital Inc, New York, USA)
Nocturnal blood oxygen saturation | baseline
  Nocturnal blood oxygen saturation (in %) will be monitored continuously during night by Nonin Wristox2 3150 (Nonin Medical Inc., Minnesota, USA)
Nocturnal blood oxygen saturation | after 12 weeks of rehabilitation
  Nocturnal blood oxygen saturation (in %) will be monitored continuously during night by Nonin Wristox2 3150 (Nonin Medical Inc., Minnesota, USA)
Breathing frequency at anaerobic threshold | baseline
  Breathing frequency (in breaths per minute) obtained during ergospirometer test using Cortex Metalyzer 3B (Cortex Biophysik GmbH, Leipzig, Germany) during a ramp protocol (starting work load of 5 Watts, increase in work load by 12.5 Watts/min).
Breathing frequency at anaerobic threshold | after 12 weeks of rehabilitation
  Breathing frequency (in breaths per minute) obtained during ergospirometer test using Cortex Metalyzer 3B (Cortex Biophysik GmbH, Leipzig, Germany) during a ramp protocol (starting work load of 5 Watts, increase in work load by 12.5 Watts/min).
Tidal volume at anaerobic threshold | baseline
  Tidal volume (in ml) obtained during ergospirometer test using Cortex Metalyzer 3B (Cortex Biophysik GmbH, Leipzig, Germany) during a ramp protocol (starting work load of 5 Watts, increase in work load by 12.5 Watts/min).
Tidal volume at anaerobic threshold | after 12 weeks of rehabilitation
  Tidal volume (in ml) obtained during ergospirometer test using Cortex Metalyzer 3B (Cortex Biophysik GmbH, Leipzig, Germany) during a ramp protocol (starting work load of 5 Watts, increase in work load by 12.5 Watts/min).
Respiratory exchange ratio at anaerobic threshold | baseline
  Respiratory exchange ratio obtained during ergospirometer test using Cortex Metalyzer 3B (Cortex Biophysik GmbH, Leipzig, Germany) during a ramp protocol (starting work load of 5 Watts, increase in work load by 12.5 Watts/min).
Respiratory exchange ratio at anaerobic threshold | after 12 weeks of rehabilitation
  Respiratory exchange ratio obtained during ergospirometer test using Cortex Metalyzer 3B (Cortex Biophysik GmbH, Leipzig, Germany) during a ramp protocol (starting work load of 5 Watts, increase in work load by 12.5 Watts/min).

SECONDARY OUTCOMES:
Functional assessment by means of the hand grip test | baseline
  Measurement of mean strength (in kg) by pulling a dynamometer handle with maximum force for 3 seconds using the dominant hand followed by 5 seconds of relaxation. Sequence in conducted 10 times.
Functional assessment by means of the hand grip test | after 12 weeks of rehabilitation
  Measurement of mean strength (in kg) by pulling a dynamometer handle with maximum force for 3 seconds using the dominant hand followed by 5 seconds of relaxation. Sequence in conducted 10 times.
Functional assessment by means of the time up and go test | baseline
  Measures the time (in s) required to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again; assesses the dynamic balance and functional mobility.
Functional assessment by means of the time up and go test | after 12 weeks of rehabilitation
  Measures the time (in s) required to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again; assesses the dynamic balance and functional mobility.
Functional assessment by means of the 6 min walking test | baseline
  Measurement of distance covered (in m) during 6 minutes of walking.
Functional assessment by means of the 6 min walking test | after 12 weeks of rehabilitation
  Measurement of distance covered (in m) during 6 minutes of walking.
Fatigue severity scale | baseline
  Questionnaire to evaluate the impact of fatigue with a minimum value of 9 (not suffering from fatigue at all) and a maximum value of 63 (highly affected by fatigue)
Fatigue severity scale | after 12 weeks of rehabilitation
  Questionnaire to evaluate the impact of fatigue with a minimum value of 9 (not suffering from fatigue at all) and a maximum value of 63 (highly affected by fatigue)
Health-related quality of life assessment by means of short form health survey (SF-36) | baseline
  Questionnaire for the assessment of health-related quality of life (minimum value = 0, low quality of life; maximum value = 100, high quality of life)
Health-related quality of life assessment by means of short form health survey (SF-36) | after 12 weeks of rehabilitation
  Questionnaire for the assessment of health-related quality of life (minimum value = 0, low quality of life; maximum value = 100, high quality of life)
Hospital Anxiety and Depression Scale | baseline
  Questionnaire for the assessment of anxiety and depression (minimum value = 0, no signs of anxiety and depression; maximum value = 10, highest levels of anxiety and depression)
Hospital Anxiety and Depression Scale | after 12 weeks of rehabilitation
  Questionnaire for the assessment of anxiety and depression (minimum value = 0, no signs of anxiety and depression; maximum value = 10, highest levels of anxiety and depression)
Bell Disability Scale | baseline
  Questionnaire for the assessment of the patient's overall functioning (minimum value = 0, worst functioning; maximum value = 100, best functioning)
Bell Disability Scale | after 12 weeks of rehabilitation
  Questionnaire for the assessment of the patient's overall functioning (minimum value = 0, worst functioning; maximum value = 100, best functioning)
Chronic Respiratory Disease Questionnaire | baseline
  Questionnaire for the assessment of dyspnoea (in post-COVID-10 patients) consisting of 5 items covering a range of 0 (worst condition) and 8 (best condition)
Chronic Respiratory Disease Questionnaire | after 12 weeks of rehabilitation
  Questionnaire for the assessment of dyspnoea (in post-COVID-10 patients) consisting of 5 items covering a range of 0 (worst condition) and 8 (best condition)
Edmonton Symptom Assessment System | baseline
  Questionnaire for the assessment of cancer symptoms consisting of 10 items covering a range of 0 (no symptoms) and 10 (worst symptoms)
Edmonton Symptom Assessment System | after 12 weeks of rehabilitation
  Questionnaire for the assessment of cancer symptoms consisting of 10 items covering a range of 0 (no symptoms) and 10 (worst symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Annaheim, Dr., Principal Investigator — Empa, Swiss Federal Laboratories for Materials Science and Technology
Locations (1):
- Klinik Gais, Gais, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
It is intended to publish the study in an open-access journal by December 2024. With this, the raw data of the physiological parameters measured and the self-reported data about fatigue symptoms (questionnaires) will be made available upon request and fulfilling the access criteria as indicated below.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available upon publication of the data Data will be available for an unlimited period of time
Access Criteria: Data will be made available upon request for scientific analysis of the data. Research objectives and data analysis plan needs to be provided.